CLINICAL TRIAL: NCT05505643
Title: COOL-IT: Cryoablation vs Lumpectomy in T1 Breast Cancers: A Randomized Controlled Trial With Safety Lead-in
Brief Title: Cryoablation vs Lumpectomy in T1 Breast Cancers
Acronym: COOL-IT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: The Foundation for Barnes-Jewish Hospital (Other); Varian Medical Systems (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202302017
Record Dates: First submitted 2022-08-15; First posted 2022-08-18 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Breast Cancer; Breast Neoplasm
Keywords: breast cancer; cryoablation; lumpectomy
MeSH Terms: conditions — Breast Neoplasms | interventions — Mastectomy, Segmental

STUDY DESIGN:
Intervention Model Description: The initial 20 participants will be enrolled to a safety lead-in arm receiving cryoablation. The next 100 participants will be randomized in a 1:1 manner to either cryoablation or lumpectomy. Patients initially treated with cryoablation who have evidence of residual or recurrent tumor on follow-up imaging will be crossed over to receive a rescue lumpectomy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (4):
- Cryoablation (Experimental): Patients will be treated with cryoablation using the Endocare SlimLine Cyroprobe under real time ultrasound guidance and local anesthesia. The cryoablation consists of a 10 minute freeze phase followed by a 10 minute passive thaw, and ends with a second 10 minute freeze cycle. The freeze-thaw-freeze times may be adjusted at the physician's discretion depending on tumor size.
  Interventions: Device: Endocare SlimLine Cryoprobe
- Lumpectomy (Active Comparator): Lumpectomy will be performed under general anesthesia as per standard operative procedures at Washington University and Siteman Cancer Center.
  Interventions: Procedure: Lumpectomy
- Rescue Arm: Lumpectomy (Other): If there is evidence of residual or recurrent tumor on follow-up imaging evaluation (6 month MRI (if can tolerate) and yearly MRI/mammography), patients in the cryoablation safety lead-in and who were randomized to receive cryoablation only will be crossed over to receive a rescue lumpectomy followed by adjuvant treatment based on standard of care.
  Interventions: Procedure: Lumpectomy
- Cryoablation - Safety Lead In (Experimental): Patients will be treated with cryoablation (Day 1) using the Endocare SlimLine Cyroprobe followed by adjuvant treatment.
  Interventions: Device: Endocare SlimLine Cryoprobe

INTERVENTIONS:
Device: Endocare SlimLine Cryoprobe — The Endocare(TM) SlimLine (TM) Cryoprobe is a single use, disposable device designed for use with Endocare Cryocare Surgical Systems. Endocare cryoprobes are designed to deliver cold temperatures for cryoablation using high-pressure argon gas circulated through the cryoprobe, followed by active thawing using helium gas.
  The Cryocare CS Surgical System is intended for use in open, minimally invasive, or endoscopic surgical procedures in the areas of general surgery, urology, gynecology, oncology, neurology, dermatology, ENT, proctology, pulmonary surgery, and thoracic surgery. The system is designed to freeze/ablate tissue by the application of extreme cold temperatures.
  Arms: Cryoablation; Cryoablation - Safety Lead In
Procedure: Lumpectomy — Patients randomized to cryoablation who experience disease recurrence may undergo crossover to lumpectomy.
  Arms: Lumpectomy; Rescue Arm: Lumpectomy

SUMMARY:
This trial studies the efficacy and safety of cryoablation in patients with low risk, early stage breast cancer. Cryoablation is a method of killing a tumor by freezing it. The standard approach for patients with this kind of cancer is a lumpectomy. This study will review the safety of the cryoablation procedure initially, followed by comparing cryoablation to lumpectomy in order to see if the cryoablation results in better disease control, complication rates, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of invasive ductal carcinoma of the breast (ER , Her-2 negative) that is grade 1 or 2 with intraductal component <25%. Must be T1N0M0 (2 cm or less).
* If DCIS is present in the biopsy specimen it should be <25% of the tumor and should be contiguous with the IDC. (i.e. DCIS should not be a separate tumor from the IDC).
* Oncotyping will be performed on T1b+Allred<6/8 and T1c tumors. Oncotype score in this subset of patients must be <26 to be included in the trial.
* At least 50 years of age.
* Mass must be visible on ultrasound and >5 mm from skin and chest wall muscles.
* Able to understand and willing to sign an IRB-approved written informed consent document.

Exclusion Criteria:

* Indication for neoadjuvant chemotherapy.
* Prior history of breast cancer.
* Breast augmentation.
* Allergy to local anesthetics.
* Pregnant or lactating. Women of childbearing potential must have a negative pregnancy test within 14 days of study entry.
* Positive axillary lymph nodes as assessed by axillary ultrasound, axillary sampling, or axillary sentinel node procedure.

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-04-03 (Actual); Primary Completion 2033-04-30 (Estimated); Study Completion 2033-04-30 (Estimated)

PRIMARY OUTCOMES:
Safety Lead-In: Number of treatment-related complications | Assessed from start of treatment through 30 days after cryoablation treatment (estimated to be 31 days)
  Excessive adverse events will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v5.0. They are defined as toxicities occurring within 30 days after the cryoablation procedure and are at least possibly related to the cryoablation. These include death, life-threatening adverse events, inpatient hospitalization or prolongation of existing hospitalization, a persistent or significant disability/incapacity, or complications related to cryoablation which interfere with adjuvant therapy such that the adjuvant therapy cannot be performed at all or delayed for a period longer than 6 months or which result in unplanned mastectomy.
Randomized Controlled Trial: Ipsilateral breast cancer recurrence (IBTR) in the treated breast. | At 5 years.
  IBTR defined from date of procedure to date of ipsilateral breast cancer recurrence, with the occurrence of ipsilateral breast tumor recurrence as the event and patients will be censored at the last follow-up.

SECONDARY OUTCOMES:
Proportion of patients who are free of serious treatment-related complications | Assessed from start of treatment through 30 days after cryoablation treatment (estimated to be 31 days)
  Excessive adverse events will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v5.0. They are defined as toxicities occurring within 30 days after the cryoablation procedure and are at least possibly related to the cryoablation. These include death, life-threatening adverse events, inpatient hospitalization or prolongation of existing hospitalization, a persistent or significant disability/incapacity, or complications related to cryoablation which interfere with adjuvant therapy such that the adjuvant therapy cannot be performed at all or delayed for a period longer than 6 months or which result in unplanned mastectomy.
Proportion of patients who demonstrate disease-free survival (DFS) | Through 5 years.
  DFS is defined as the time from procedure to time of ipsilateral recurrence, contralateral recurrence, regional recurrence or distant metastasis, or date of last follow-up if none of the recurrence events occur.
Overall survival (OS) | Through 5 years.
  OS is defined from date of procedure to date of death or date of last follow up if none of the recurrence events occur.

CONTACTS AND LOCATIONS:
Overall Officials: Heather Garrett, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the de-identified individual participant data and the study protocol will be made available to investigators who provide a methodologically sound proposal. Proposals should be directed to hvgarrett@wustl.edu. De- identified individual participant data will also be made available to Varian.
Supporting Information: Study Protocol, SAP
Access Criteria: Proposals should be directed to hvgarrett@wustl.edu.

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu